CLINICAL TRIAL: NCT06266572
Title: Overcoming Stigma and Improving Outcomes for SUDs Through Education, Engagement,
Brief Title: Overcoming Stigma and Improving Outcomes for SUDs Through Education, Engagement, and Empowerment
Acronym: OASIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R43DA055182-01 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention (Experimental): Research participants will receive access to a web-based platform designed to provide information about Opioid Use Disorder. Prior to receiving access to this application, research participants will complete online, self-reported surveys assessing stigma, empowerment, and knowledge of opioids.
  Interventions: Behavioral: Overcoming and Addressing Stigma in Substance Use Disorders (OASIS)
- Post-Intervention (Experimental): Research participants will have access to the web-based platform for 7 to 14 days prior to receiving a second, identical series of self-report surveys assessing stigma, empowerment, and knowledge of opioids. Additionally, after using the platform, research participants will complete a measure of system usability.
  Interventions: Behavioral: Overcoming and Addressing Stigma in Substance Use Disorders (OASIS)

INTERVENTIONS:
Behavioral: Overcoming and Addressing Stigma in Substance Use Disorders (OASIS) — Web-based educational platform for clinicians and individuals with OUD that will decrease barriers to care and enhance treatment outcomes

SUMMARY:
C4 Innovations (C4) and partners at Yale University (Yale) and the West Haven VA Medical Center (WHVA) proposed to develop and test OASIS (Overcoming and Addressing Stigma in Substance Use Disorders), a web-based educational platform for primary care clinicians and individuals with Opioid Use Disorder. The major aims of the study were to:

1. Develop a prototype of OASIS for patients with Opioid Use Disorder (OUD) and primary care clinicians; conduct usability testing.
2. Pilot OASIS with a small sample of individuals with untreated OUD and their clinicians to determine feasibility, acceptability, and preliminary product effectiveness for a Phase II effectiveness trial.

After development of the prototype, the C4-Yale-WHVA team planned to test OASIS with patients (N = 30) and clinicians (N = 5) using validated measures and qualitative interviews to assess usability, satisfaction, knowledge, empowerment, and stigma.

ELIGIBILITY:
Inclusion Criteria:

For providers:

* Clinically active and seeing patients;
* Having a device with Internet access to use the OASIS prototype
* English speaking
* Willing and able to complete data collection activities.

For patients:

* Diagnosed OUD
* Unmet substance use treatment need
* Has an upcoming primary care visit scheduled for the intervention period (1-2 months)
* English speaking
* Has access to a device with Internet access to use the OASIS prototype
* Willing and able to complete data collection activities

Exclusion Criteria:

Patient participants will be excluded from this study if they:

1) Currently receiving or have received medication for opioid dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Open Minds Scale for Health Care Providers | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  Description: A 20-item scale assessing stigma in health care providers, rated on a 5 point likert scale from Strongly Disagree (1) to Strongly Agree (5).
Brief Opioid Stigma Scale | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  An 8-item scale assessing perceptions of stigma and endorsed stigma toward individuals using opioids. Rated on a 5 point likert scale from Strongly Disagree (1) to Strongly Agree (5). Providers in this study did not complete the items on the Harm subscale, items 9-12.
Perceived Stigma of Addiction Scale | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  An 8-item scale assessing perceptions of stigma towards individuals with substance use disorders. Rated on a 7 point likert scale from Very Strongly Disagree (1) to Very Strongly Agree (7).
Knowledge Check | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week
  A 10-item assessment developed by the research team to assess knowledge of opioids and opioid use disorder
System Usability Scale | Assess only at the post-assessment, after using the platform for at least one week.
  A 10-item measure assessing the overall usability of the online platform. Rated on a 5 point likert scale from Strongly Disagree (1) to Strongly Agree (5).
Internalized Stigma of Mental Illness Scale | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  A 29-item measure assessing the participant's own stigma relating to mental illness. Rated on a 4 point likert scale from Strongly Disagree (1) to Strongly Agree (4).
Recovery Empowerment Scale | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  A 20-item scale assessing a participant's levels of empowerment, rated on a 7 point likert scale from Almost Never (1) to Almost Always (7).
Mental Health Seeking Attitudes Scale | Assessed at both timepoints: prior to accessing the online platform and after using the platform for at least one week.
  A 9-item scale assessing the individuals rating between two dichotomous choices and how accurately they describe their perceptions of help-seeking. Participants are asked to choose one of two words on a scale (e.g., useless vs. useful) and are asked to rate how strongly they feel this word describes their thoughts on a scale from Undecided (0) to Extremely (3).

CONTACTS AND LOCATIONS:
Locations (1):
- West Haven VA Medical Center, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No